CLINICAL TRIAL: NCT06872944
Title: Effect of Melatonin on Postoperative Pain After Simple Nephrectomy: A Randomized Double-Blinded Controlled Study
Brief Title: Effect of Melatonin on Postoperative Pain After Simple Nephrectomy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Karim Hussein, lecturer of anesthesia-faculty of medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: melatonin in nephrectomy
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Pain Score (VAS) at 24 h Postoperatively
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M (Experimental): Patients will receive 4 mg of prolonged-release formulation of oral melatonin at the night (8 PM) before the procedure and another dose 2 hours before surgery.
  Interventions: Drug: Melatonin
- Group C (Placebo Comparator): Patients will receive sugar coated tablets at the night (8 PM) before the procedure and another dose 2 hours before surgery.
  Interventions: Drug: Sugar Coated Tablet

INTERVENTIONS:
Drug: Melatonin — Melatonin, or N-acetylmethoxytryptamine, is a hormone secreted by the pineal gland in the brain. Light is the main factor that regulates melatonin production. Melatonin has important biological effects on the body and plays an important role in regulating the sleep wake cycle. Besides circadian rhythm stabilizing, exogenous melatonin has been investigated for other effects such as modulation of blood pressure, body temperature and cortisol control, immune function, and anti-oxidative defense.
  Recent studies showed some benefits of perioperative short-acting melatonin in different groups of patients such as quality of recovery after surgery, diminished depressive symptoms and pain score reduction
  Arms: Group M
Drug: Sugar Coated Tablet — sugar coated tablets will be given to the patients at the night (8 PM) before the procedure and another dose 2 hours before surgery
  Other Names: placebo
  Arms: Group C

SUMMARY:
The aim of the study is to evaluate the role of melatonin in the management of postoperative pain in patients undergoing simple nephrectomy regarding:

* Pain score (VAS).
* Total Morphine consumption is 1st 24 hr.
* Time to the 1st rescue analgesia.
* Intra-operative and post-operative hemodynamics.
* Anxiety.
* Patient satisfaction.
* Adverse events.

DETAILED DESCRIPTION:
This study will be conducted in Cairo University Hospitals at Uorolgy OR. This study will include 40 patients divided into two groups, aged 18 to 65 years, both sexes, belonging to the American Society of Anesthesiologists (ASA) physical status I, II undergoing simple nephrectomy.

1. Inclusion criteria

   * Age from 18 to 65 years.
   * Both sexes.
   * (ASA) physical status I, II.
   * Patients undergoing simple nephrectomy.
2. Exclusion criteria

   * Patient refusal.
   * Patients with a history of allergic reactions to melatonin.
   * Patients receiving drugs with known analgesic and sedative properties.
   * Body Mass Index (BMI) over 30 kg/m2.
   * Drug or alcohol abuse.
   * History of cardiovascular disease.
   * Renal Failure.
   * Mental impairment.
   * Renal impairment.

Medical and surgical history of the patients will be taken, clinical examination of the patients will be performed and routine laboratory investigations as CBC, coagulation studies, renal function and liver function will be done.

Preoperative visit will be conducted the day before surgery. All patients will be evaluated by the same anesthesia resident, who provided information on the preoperative course and instructed them on the procedure.

Each patient will be instructed about postoperative pain assessment with the visual analog scale (VAS) which [0 represents "no pain" while 10 represents "the worst pain imaginable"] and level of anxiety.

Intraoperative management All patients will be connected to standard monitoring which include electrocardiography (ECG), non-invasive arterial blood pressure (NIBP), pulse oximetry, temperature probe, and capnography (will be connected after induction of general anesthesia).

Induction of general anesthesia will be done after inserting 20G venous cannula by IV propofol 2-2.5 mg / kg and IV fentanyl 2ug / kg. After IV Atracurium 0.5mg / kg, endotracheal intubation will be done.

Maintenance of anesthesia will be isoflurane (1-1.5%) with 50-100% oxygen. Incremental doses of IV Atracurium 0.1mg/Kg will be given every 20 min. Patients will be mechanically ventilated and end-tidal CO2 will be maintained between 35-45 mmHg.

Additional fentanyl bolus dosages of 1 µg/kg IV will be administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline (after exclusion of other causes than pain).

At the end of the surgery, inhalational anesthetics will be stopped waiting for motor power and conscious level to be regained. Then the reversal will be given IV Neostigmine 0.03-0.07 mg/kg + Atropine 0.02 mg/kg.

A standardized analgesic regimen will be prescribed in the post-operative period. All patients will receive paracetamol 1 gm every 6 h as routine analgesia.

Rescue analgesia of morphine will be given as 3 mg bolus if the VAS > 3 to be repeated after 30 min if pain persists until the VAS < 4. VAS will be assessed at 0, 2, 4, 6, 8, 12, 18, and 24 h postoperatively. The adverse effects will be assessed: hypotension (decrease in basal mean arterial blood pressure by 20%) will be treated with I.V. fluid, bradycardia (defined by decrease in basal heart rate by 20%) will be treated by I.V. atropine 0.02 mg/kg, respiratory depression (the SpO2 < 95% and need O2 supplementation), and 4 mg of ondansetron every 6 hours will be administered for postoperative nausea/vomiting (PONV) as required.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* (ASA) physical status I, II.
* Patients undergoing simple nephrectomy.

Exclusion Criteria:

* Patient refusal.

  * Patients with a history of allergic reactions to melatonin.
  * Patients receiving drugs with known analgesic and sedative properties.
  * Body Mass Index (BMI) over 30 kg/m2.
  * Drug or alcohol abuse.
  * History of cardiovascular disease.
  * Renal Failure.
  * Mental impairment.
  * Renal impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-06-21 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Pain score (VAS) at 24 h postoperatively | 24 hours postoperative
  A standardized analgesic regimen will be prescribed in the post-operative period. All patients will receive paracetamol 1 gm every 6 h as routine analgesia.
  Rescue analgesia of morphine will be given as 3 mg bolus if the VAS > 3 to be repeated after 30 min if pain persists until the VAS < 4. VAS will be assessed at 0, 2, 4, 6, 8, 12, 18, and 24 h postoperatively.

SECONDARY OUTCOMES:
Time to the 1st rescue analgesia | (time from end of surgery to first dose of morphine administrated 24 hours postoperative.
  (time passed from end of the surgery till the patient require the first dose of morphine
Total Morphine consumption is 1st 24 hr (mg). | 24 hours postoperative
  total amount of morphine consumed by the patient in first 24 hours postoperative
Degree of patient satisfaction | 24 hours postoperative
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied)

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Medicine-Cairo Univeristy, Cairo
  - Faculty of Medicine- Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bonmati-Carrion MA, Rol MA. Melatonin as a Mediator of the Gut Microbiota-Host Interaction: Implications for Health and Disease. Antioxidants (Basel). 2023 Dec 23;13(1):34. doi: 10.3390/antiox13010034. PMID 38247459
- [Background] Kiabi FH, Emadi SA, Jamkhaneh AE, Aezzi G, Ahmadi NS. Effects of preoperative melatonin on postoperative pain following cesarean section: A randomized clinical trial. Ann Med Surg (Lond). 2021 May 12;66:102345. doi: 10.1016/j.amsu.2021.102345. eCollection 2021 Jun. PMID 34040762
- [Background] Andersen LP. The analgesic effects of exogenous melatonin in humans. Dan Med J. 2016 Oct;63(10):B5289. PMID 27697139
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] Chen Q, Beal EW, Okunrintemi V, Cerier E, Paredes A, Sun S, Olsen G, Pawlik TM. The Association Between Patient Satisfaction and Patient-Reported Health Outcomes. J Patient Exp. 2019 Sep;6(3):201-209. doi: 10.1177/2374373518795414. Epub 2018 Aug 27. PMID 31535008